CLINICAL TRIAL: NCT02691286
Title: Prognostic Value of Circulating microRNAs in Patients With ST-elevation Myocardial Infarction (STEMI) Complicated by Cardiogenic Shock
Brief Title: Circulating microRNAs in Patients With STEMI Complicated With Cardiogenic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-RNA-2015-80
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: STEMI; Cardiogenic Shock; Acute Coronary Syndrome; microRNA
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Shock, Cardiogenic; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA and LiHe tubes with 10 ml of blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cardiogenic Shock STEMI: Patients admitted to the hospital with the diagnosis with STEMI complicated with cardiogenic shock
- No Cardiogenic Shock STEMI: Patients admitted to the hospital with the diagnosis with STEMI without cardiogenic shock

SUMMARY:
The aim of the study is knowing the prognostic value of circulating miRNAs in patients admitted to our hospital with STEMI complicated with cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ST elevation by ECG diagnostic of STEMI
* Evidency of coronary occlusion in coronariography
* Signed informed consent

Exclusion Criteria:

* Patients admitted from other hospitals
* Impossibility of getting blood samples in first 6h
* Declined consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Hospital de la Santa Creu i Sant Pau with diagnosis of STEMI with or without cardiogenic shock
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-08 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sans-Roselló, M.D., Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No